CLINICAL TRIAL: NCT03444948
Title: A Phase II Prospective Randomised Clinical Study of Endoscopic Ultrasound Guided Radiofrequency Ablation (EUS-RFA) for Inoperable Pancreatic Ductal Adenocarcinoma
Brief Title: A Clinical Study of EUS-RFA for Inoperable Pancreatic Ductal Adenocarcinoma
Acronym: EUS-RFA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: There was a voluntary recall from the Habib EUS RFA device manufacturer
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE 17.215; NCT03065985 (obsolete NCT alias)
Record Dates: First submitted 2017-10-27; First posted 2018-02-26 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3 radiofrequency ablation procedures (Experimental): Subject will undergo 3 radiofrequency ablation procedures at 1 month intervals (EUS-RFA using Habib Tm as a probe)
  Interventions: Device: EUS-RFA using Habib Tm as a probe
- standard medical care (Active Comparator): Subject will receive standard medical care, including pain relief drugs
  Interventions: Procedure: EUS

INTERVENTIONS:
Device: EUS-RFA using Habib Tm as a probe — 3 EUS-RFA interventions at 1-month interval
  Arms: 3 radiofrequency ablation procedures
Procedure: EUS — Standard intervention
  Arms: standard medical care

SUMMARY:
To assess if endoscopic ultrasound-guided radiofrequency ablation application in patients with inoperable pancreatic cancer confers survival benefit when compared to patients receiving standard medical care.

DETAILED DESCRIPTION:
The five-year survival for pancreatic ductal adenocarcinoma (PDAC) is less than 5% in spite of the advances in management of cancers in the last few decades. Endobiliary application of radiofrequency (RF) has been developed and used in patients with inoperable bile duct and pancreatic head adenocarcinomas presenting with biliary obstruction. (1, 2) Endoscopic ultrasound (EUS) radiofrequency ablation (RFA) of pancreatic neoplasms has been proven to be well tolerated and safe, inducing a significant reduction in tumour size (3). Various techniques of EUS-guided tumour ablation have been described, including RF ablation, photodynamic therapy, laser ablation, and ethanol injection (4). Kahaleh et al. have demonstrated that Endoscopic ultrasound guided RF ablation (EUS-RFA) of the pancreatic head using Habib EUS-RFA catheter (EMcision Ltd, UK) through a 19-gauge needle was well tolerated in 5 Yucatan pigs and with minimum amount of pancreatitis (5). In a pilot clinical study, Pai et al showed either a complete response or at least a 50% reduction in tumours following application of radiofrequency ablation with the Habib™ EUS-RFA device in a group of eight patients with pancreatic cancers (3).

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age.
* A cytological / histological diagnosis of inoperable PDAC based on multidisciplinary review of cross-sectional imaging and cytology / histology results.
* Patients ought to be fit enough to be considered for the study (ECOG (Eastern Cooperative Oncology Group) performance status 0, 1 or 2)
* Patients who have commenced chemotherapy are not excluded from the study
* Patients capable of giving informed consent
* Negative blood pregnancy test for women of childbearing potential
* Willingness and ability to comply with all protocol requirements including scheduled visits, treatment plans, laboratory tests and other study procedures.

Exclusion Criteria:

* ECOG performance status 3 or 4
* Life expectancy less than 3 months (including liver metastases, carcinomatosis)
* Prior investigational drugs within the last 30 days
* Known infection with human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 1 month
  Duration of survival
Survival | at time of death on average 10months
  Duration of survival

SECONDARY OUTCOMES:
Quality of life (HEALTH, SOCIAL INTERACTIONS, DAILY ACTIVITIES) | 1 month
  Quality of life questionnaire DDQ15
Quality of life (HEALTH, SOCIAL INTERACTIONS, DAILY ACTIVITIES) | Time of death on average 10 months
  Quality of life questionnaire DDQ15
Pain reduction | 1 month
  Likert Scale
Pain reduction | Time of death on average 10months
  Likert Scale
Tumour Size | 4 months
  Measures during follow-upEUS
Monitoring of Adverse reactions | At time of death on average 10months
  Number of participants with treatment-related adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: ANAND V SAHAI, MD, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (1):
- Centre de recherche du Centre hospitalier de l'université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No